CLINICAL TRIAL: NCT01604018
Title: An Optional Two Year Follow Up Study to Evaluate the Continued Efficacy of Cat-PAD ToleroMune Peptide Immunotherapy in Cat Allergic Subjects Following Challenge to Cat Allergen in an Environmental Exposure Chamber
Brief Title: An Optional Two Year Follow Up Study to Study CP005A
Status: Completed | Type: Observational
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Cetero Research, Toronto (Unknown)
Responsible Party: Sponsor
Other Study IDs: CP005B
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Cat Allergy; Rhinoconjunctivitis
Keywords: Cat Allergy; Rhinoconjunctivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Placebo: Subjects previously randomized to receive placebo in study CP005 and completed CP005A.
- Cat-PAD Group 1: Subjects previously randomized to receive Cat-PAD dose 1 in study CP005 and completed CP005A.
- Cat-Pad Group 2: Subjects previously randomized to receive Cat-PAD dose 2 in study CP005 and completed CP005A.

SUMMARY:
Cat allergy is an increasingly prevalent condition affecting 10-15% of patients with allergic rhinoconjunctivitis and/or asthma.

The purpose of this optional observational follow-on study is to further evaluate rhinoconjunctivitis symptoms on exposure to cat dander in the EEC among subjects who completed all dosing visits in study CP005 and all visits in study CP005A approximately two years after the start of treatment.

DETAILED DESCRIPTION:
Subjects who completed all visits in studies CP005 and CP005A will be invited to attend the Screening Visit for CP005B. Subjects will attend for 4 visits to the EEC on successive days. Following the last EEC visit is a follow-up visit which will be performed 3-10 days later.

ELIGIBILITY:
Inclusion Criteria:

- Previously randomised into study CP005 and completed all visits in the follow-on study CP005A

Exclusion Criteria:

* "Partly controlled" and "uncontrolled" asthma
* History of anaphylaxis to cat allergen
* Subjects with an FEV1 < 70% of predicted
* Subjects who cannot tolerate baseline challenge in the EEC
* Treatment with beta-blockers, alpha-adrenoceptor blockers, tranquilizers, or psychoactive drugs
* Symptoms of a clinically relevant illness, in the Investigator's opinion, within 6 weeks prior to Screening Visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects previously randomised in study CP005 and completed all dosing and PTC in CP005 and all visits in CP005A.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Total Rhinoconjunctivitis Symptom Score | 102-106 weeks after the start of treatment in CP005

SECONDARY OUTCOMES:
Total Symptom scores for ocular and nasal symptoms | 102-106 weeks after the start of treatment in CP005

CONTACTS AND LOCATIONS:
Overall Officials: Peter Couroux, MD, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada